CLINICAL TRIAL: NCT06268886
Title: A Randomized, Double-blind, Placebo-controlled, Global Proof-of-concept Study to Evaluate the Efficacy, Safety, and Tolerability of BMS-986446, an Anti-MTBR Tau Monoclonal Antibody, in Participants With Early Alzheimer's Disease (TargetTau-1)
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of an Anti-MTBR Tau Monoclonal Antibody (BMS-986446) in Participants With Early Alzheimer's Disease
Acronym: TargetTau-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN008-0003; 2023-504840-32 (Other: EU CTR); U1111-1290-3539 (Registry Identifier: WHO)
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Alzheimer Disease; BMS-986446; Neurodegenerative disease; Dementia; Brain Diseases; Anti-MTBR tau monoclonal antibody; TargetTau-1; Anti-tau therapy
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases; Dementia; Brain Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- BMS-986446 Dose A (Experimental)
  Interventions: Drug: BMS-986446
- BMS-986446 Dose B (Experimental)
  Interventions: Drug: BMS-986446

INTERVENTIONS:
Drug: BMS-986446 — Specified dose on specified days
  Arms: BMS-986446 Dose A; BMS-986446 Dose B
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness, safety, and tolerability of BMS-986446 an Anti-MTBR Tau Monoclonal Antibody in participants with Early Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria

* Mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or mild AD dementia consistent with the National Institute on Aging and the Alzheimer's Association (NIA-AA) core clinical criteria.
* Global Clinical Dementia Rating (CDR) score of 0.5 to 1.0 and a CDR-Memory Box score of 0.5 and greater at screening and Baseline.
* Evidence of AD pathology.
* Objective impairment in episodic memory as indicated by at least 1 standard deviation below age-adjusted mean in the Wechsler Memory Scale IV-Logical Memory Subtest II (WMS-IV LM II).
* Mini Mental Status Examination (MMSE) score ≥ 20 to 28 (inclusive).

Exclusion Criteria

* Any evidence of a condition that may affect cognition other than AD.
* Contraindications to PET imaging.
* Inability to tolerate or contraindication to magnetic resonance imaging.
* Any serious medical condition that could, in the opinion of the investigator, affect the participant's safety or interfere with study assessments.
* Geriatric Depression Scale (GDS) score greater than or equal to 8 at screening.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-03-18 (Estimated); Study Completion 2027-03-18 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in brain tau deposition as measured by tau positron emission tomography (PET) | At week 76

SECONDARY OUTCOMES:
Change from baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) score | At week 76
Change from baseline in integrated Alzheimer's Disease Rating Scale (iADRS) score | At week 76
Change from baseline in Alzheimer's Disease Assessment Scale-Cognitive subscale (ADASCog14) score | At week 76
Change from baseline in Alzheimer's Disease Cooperative Study-instrumental Activities of Daily Living scale (ADCS-iADL) score | At week 76
Change from baseline in Mini Mental State Examination (MMSE) score | At week 76

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (176):
- United States (119):
  - Local Institution - 0068, Chandler, Arizona
  - Local Institution - 0102, Gilbert, Arizona
  - Local Institution - 0019, Phoenix, Arizona
  - Local Institution - 0018, Scottsdale, Arizona
  - Local Institution - 0026, Scottsdale, Arizona
  - Local Institution - 0077, Tucson, Arizona
  - Local Institution - 0038, Tucson, Arizona
  - Local Institution - 0164, Encino, California
  - Local Institution - 0139, Fullerton, California
  - Local Institution - 0191, Irvine, California
  - Local Institution - 0234, Long Beach, California
  - Local Institution - 0142, Los Alamitos, California
  - Local Institution - 0037, Napa, California
  - Local Institution - 0209, Sacramento, California
  - Local Institution - 0052, San Francisco, California
  - Local Institution - 0137, Santa Ana, California
  - Local Institution - 0046, Sherman Oaks, California
  - Local Institution - 0106, Danbury, Connecticut
  - Local Institution - 0148, New Haven, Connecticut
  - Local Institution - 0056, New Haven, Connecticut
  - Local Institution - 0153, Stamford, Connecticut
  - Local Institution - 0022, Altamonte Springs, Florida
  - Local Institution - 0048, Atlantis, Florida
  - Local Institution - 0228, Boca Raton, Florida
  - Local Institution - 0250, Boca Raton, Florida
  - Local Institution - 0224, Bradenton, Florida
  - Local Institution - 0020, Clermont, Florida
  - Local Institution - 0009, Daytona Beach, Florida
  - Local Institution - 0213, Fort Myers, Florida
  - Local Institution - 0059, Greenacres City, Florida
  - Local Institution - 0207, Hialeah, Florida
  - Local Institution - 0212, Hialeah, Florida
  - Local Institution - 0198, Hialeah, Florida
  - Local Institution - 0151, Lady Lake, Florida
  - Local Institution - 0146, Lakeland, Florida
  - Local Institution - 0192, Maitland, Florida
  - Local Institution - 0143, Maitland, Florida
  - Local Institution - 0027, Merritt Island, Florida
  - Local Institution - 0203, Miami, Florida
  - Local Institution - 0058, Miami, Florida
  - Local Institution - 0034, Miami, Florida
  - Local Institution - 0211, Miami, Florida
  - Local Institution - 0195, Miami, Florida
  - Local Institution - 0014, Miami, Florida
  - Local Institution - 0005, Miami, Florida
  - Local Institution - 0208, Miami, Florida
  - Local Institution - 0013, Miami, Florida
  - Local Institution - 0008, Miami, Florida
  - Local Institution - 0199, Miami, Florida
  - Local Institution - 0206, Miami, Florida
  - Local Institution - 0176, Miami, Florida
  - Local Institution - 0071, Miami, Florida
  - Local Institution - 0156, Miami, Florida
  - Local Institution - 0249, Miami, Florida
  - Local Institution - 0039, Miami, Florida
  - Local Institution - 0225, Miami, Florida
  - Local Institution - 0197, Miami Springs, Florida
  - Local Institution - 0217, Naples, Florida
  - Local Institution - 0017, New Port Richey, Florida
  - Local Institution - 0144, Ocala, Florida
  - Local Institution - 0202, Orlando, Florida
  - Local Institution - 0219, Orlando, Florida
  - Local Institution - 0035, Orlando, Florida
  - Local Institution - 0238, Orlando, Florida
  - Local Institution - 0210, Port Orange, Florida
  - Local Institution - 0204, Sarasota, Florida
  - Local Institution - 0012, Stuart, Florida
  - Local Institution - 0136, Stuart, Florida
  - Local Institution - 0200, Tampa, Florida
  - Local Institution - 0080, Tampa, Florida
  - Local Institution - 0087, Tampa, Florida
  - Local Institution - 0042, Tampa, Florida
  - Local Institution - 0194, Viera, Florida
  - Local Institution - 0011, Wellington, Florida
  - Local Institution - 0223, West Palm Beach, Florida
  - Local Institution - 0149, West Palm Beach, Florida
  - Local Institution - 0029, Windermere, Florida
  - Local Institution - 0101, Winter Park, Florida
  - Local Institution - 0154, Winter Park, Florida
  - Local Institution - 0105, Columbus, Georgia
  - Local Institution - 0236, Chicago, Illinois
  - Local Institution - 0021, Chicago, Illinois
  - Local Institution - 0161, Elk Grove Village, Illinois
  - Local Institution - 0003, Gurnee, Illinois
  - Local Institution - 0145, Park Ridge, Illinois
  - Local Institution - 0081, Springfield, Illinois
  - Local Institution - 0235, Boston, Massachusetts
  - Local Institution - 0025, Boston, Massachusetts
  - Local Institution - 0015, Braintree, Massachusetts
  - Local Institution - 0174, Foxborough, Massachusetts
  - Local Institution - 0118, Methuen, Massachusetts
  - Local Institution - 0040, Newton, Massachusetts
  - Local Institution - 0120, Plymouth, Massachusetts
  - Local Institution - 0045, Watertown, Massachusetts
  - Local Institution - 0119, Portsmouth, New Hampshire
  - Local Institution - 0031, Princeton, New Jersey
  - Local Institution - 0062, Toms River, New Jersey
  - Local Institution - 0060, Albany, New York
  - Local Institution - 0157, Amherst, New York
  - Local Institution - 0061, Manhasset, New York
  - Local Institution - 0205, New York, New York
  - Local Institution - 0214, New York, New York
  - Local Institution - 0104, New York, New York
  - Local Institution - 0133, New York, New York
  - Local Institution - 0043, Matthews, North Carolina
  - Local Institution - 0215, Dayton, Ohio
  - Local Institution - 0155, Independence, Ohio
  - Local Institution - 0023, Plymouth Meeting, Pennsylvania
  - Local Institution - 0024, East Providence, Rhode Island
  - Local Institution - 0163, Providence, Rhode Island
  - Local Institution - 0132, Cordova, Tennessee
  - Local Institution - 0140, Franklin, Tennessee
  - Local Institution - 0222, Nashville, Tennessee
  - Local Institution - 0069, Austin, Texas
  - Local Institution - 0033, Beaumont, Texas
  - Local Institution - 0051, Dallas, Texas
  - Local Institution - 0016, Houston, Texas
  - Local Institution - 0196, Fairfax, Virginia
  - Local Institution - 0168, Richmond, Virginia
- Australia (9):
  - Local Institution - 0111, East Gosford, New South Wales
  - Local Institution - 0170, Macquarie Park, New South Wales
  - Local Institution - 0116, Griffith University, Queensland
  - Local Institution - 0115, Carlton North, Victoria
  - Local Institution - 0093, Ivanhoe, Victoria
  - Local Institution - 0001, Malvern, Victoria
  - Local Institution - 0125, Melbourne, Victoria
  - Local Institution - 0147, Parkville, Victoria
  - Local Institution - 0094, Nedlands, Western Australia
- Belgium (5):
  - Local Institution - 0122, Anderlecht, Brussels Capital
  - Local Institution - 0175, Antwerpen, Brussels Capital
  - Local Institution - 0082, Kortrijk, VWV
  - Local Institution - 0097, Brussels
  - Local Institution - 0076, Leuven
- Canada (7):
  - Local Institution - 0112, Ottawa, Ontario
  - Local Institution - 0047, Toronto, Ontario
  - Local Institution - 0044, Toronto, Ontario
  - Local Institution - 0109, Toronto, Ontario
  - Local Institution - 0113, Greenfield Park, Quebec
  - Local Institution - 0248, Montreal, Quebec
  - Local Institution - 0053, Québec
- Japan (20):
  - Local Institution - 0181, Nagoya, Aichi-ken
  - Local Institution - 0227, Toride-Shi, Ibaraki
  - Local Institution - 0186, Kurashiki-Shi, Okayama-ken
  - Local Institution - 0242, Hirakata-Shi, Osaka
  - Local Institution - 0253, Osaka, Osaka
  - Local Institution - 0185, Bunkyo-Ku, Tokyo
  - Local Institution - 0218, Hachioji-Shi, Tokyo
  - Local Institution - 0184, Setagaya-Ku, Tokyo
  - Local Institution - 0226, Chūōku
  - Local Institution - 0190, Himeji-shi
  - Local Institution - 0188, Kasukabe-Shi
  - Local Institution - 0179, Kodaira-Shi
  - Local Institution - 0221, Musashimurayama-Shi
  - Local Institution - 0220, Musashino-shi
  - Local Institution - 0180, Nagoya
  - Local Institution - 0178, Osaka
  - Local Institution - 0232, Ōbu
  - Local Institution - 0240, Tachikawa-Shi
  - Local Institution - 0239, Takatsuki-Shi
  - Local Institution - 0189, Toyonaka-Shi
- Local Institution - 0091, Singapore, Singapore
- South Korea (4):
  - Local Institution - 0117, Songpa-gu, Seoul
  - Local Institution - 0110, Gwangjingu
  - Local Institution - 0050, Incheon
  - Local Institution - 0114, Junggu
- Spain (6):
  - Local Institution - 0158, Barcelona, B
  - Local Institution - 0054, Sant Cugat del Vallès, CT
  - Local Institution - 0231, Lleida, L
  - Local Institution - 0096, Barcelona
  - Local Institution - 0171, Barcelona
  - Local Institution - 0172, Barcelona
- Local Institution - 0167, Malmo, M, Sweden
- United Kingdom (4):
  - Local Institution - 0121, Enfield, LND
  - Local Institution - 0252, London, LND
  - Local Institution - 0247, Bath, SOM
  - Local Institution - 0089, Chertsey, Surrey

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06268886.html